CLINICAL TRIAL: NCT03773328
Title: Phase I Trial To Evaluate The Safety Of CK0801 In Treatment-Resistant Guillain-Barré Syndrome (GBS)
Brief Title: A Clinical Trial of CK0801 (a New Drug) In Patients With Treatment-Resistant Guillain-Barré Syndrome (GBS)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Pending contract negotiations
Sponsor: Cellenkos, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CK0801-201-1
Record Dates: First submitted 2018-10-23; First posted 2018-12-12 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Guillain-Barré Syndrome
MeSH Terms: conditions — Guillain-Barre Syndrome

STUDY DESIGN:
Intervention Model Description: Open-label, single arm study using a Simon 3 + 3 design. Study will utilize 3 dose cohorts with a minimum of 3 patients in each cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CK0801, 50ml (Experimental): All subjects will receive adoptive therapy with an infusion of unrelated cord blood-derived regulatory T cells: CK0801. Subjects will receive one 50mL intravenous dose of CK0801 (Treg cells) on study Day 0. A total of three cohorts will be evaluated.
  Cohort dosing will be as follows:
  Dose level 1 = 1x10e6/kg Treg cells per kg recipient ideal body weight (IBW); Dose level 2 = 3x10e6/kg Treg cells per kg recipient ideal body weight (IBW); Dose level 3 = 1x10e7/kg Treg cells per kg recipient ideal body weight (IBW).
  Interventions: Biological: CK0801

INTERVENTIONS:
Biological: CK0801 — CK0801 (Cord blood-derived T-regulatory cells)

SUMMARY:
The goal of this research study is to determine whether it is safe and practical to give CK0801 (a cord-blood derived T-regulatory cell product) to patients with Guillain-Barré Syndrome (GBS). Researchers also want to determine the highest possible dose that is safe to be given and to learn if CK0801 may improve the symptoms of GBS. There will be three doses of CK0801 given during this study. A minimum of three patients will be treated in each dose level. The dose a patient receives is dependent on the timing of when they enter the study, as after each dose level is completed the following patients will receive the next highest dose level.

DETAILED DESCRIPTION:
CK0801 (Cord blood-derived T-regulatory cells) consists of ex vivo expanded T-regulatory cells with a flow cytometry phenotype of ≥ 60% CD4+CD25+ T-regulatory (Treg) cells and < 10% CD4-CD8+ T-cytotoxic/suppressor cells. The cellular starting material of CK0801 is a single unit of umbilical cord blood (CBU) from a normal, healthy unrelated donor. Because Treg cells are present only at low frequency in circulating blood or umbilical cord blood, production of clinically relevant Treg cell doses requires ex vivo enrichment and expansion of Treg cells with a CD4+CD25+ phenotype. In their natural state, T-regulatory (Treg) cells play an important role in maintaining immune homeostasis and limiting autoimmune responses by modulating both innate and adaptive immunity. Based on literature reports of animal studies showing induction of immune tolerance by Treg cells in autoimmune diseases, graft-versus-host disease, and solid organ transplant rejection, the administration of Treg cells in human clinical trials has become an attractive strategy to induce immune tolerance in patients in a variety of clinical settings.

ELIGIBILITY:
Inclusion Criteria:

1. Subject fulfills the diagnostic criteria for Guillain-Barré syndrome (GBS) (Appendix 1).
2. HLA matched (≥ 3/6 at HLA-A, HLA-B, and HLA-DRB1) cord blood unit available for CK0801 generation.
3. Subjects age 18 to 70 years.
4. Subject has GBS disability scale score of 4 and unchanged 1 week after IVIG or PE treatment (Appendix 2).
5. Subject has completed IVIG/PE treatment ≥ 4 weeks prior to CK0801 infusion.
6. Subject has modified Erasmus GBS outcome score (mEGOS score) of ≥7 at the time of presentation and unchanged 1 week after IVIG or PE treatment (Table 3).
7. Bilirubin ≤ 2 x ULN and, ALT ≤ 2 x ULN (unless Gilbert's syndrome).
8. Calculated creatinine clearance of > 50mL/min using the Cockroft-Gault equation for adult patients 18 - 70 years old.
9. Female subjects of child bearing potential (FPCP) must have a negative urine or serum pregnancy test. NOTE: FPCP is defined as premenopausal and not surgically sterilized. FPCP must agree to use maximally effective birth control or to abstain from heterosexual activity throughout the study. Effective contraceptive methods include intra-uterine device, oral and/or injectable hormonal; contraception, or 2 adequate barrier methods (e.g., cervical cap with spermicide, diaphragm with spermicide).
10. Subject has agreed to abide by all protocol required procedures including study-related assessments, visits and long term follow up.
11. Subject is willing and able to provide written informed consent. If subject is temporarily unable to sign the consent due to disease-related complications (e.g., upper extremity paralysis), a legally authorized representative (LAR) will be used. The subject will sign the consent as soon as they are capable.

Exclusion Criteria:

1. Subject has received immunotherapy, chemotherapy, biologic or investigational agent within 4 weeks prior to CK0801 infusion.
2. Subject has received prior CB Treg therapy.
3. Subject has uncontrolled infection, not responding to appropriate antimicrobial agents after seven days of therapy. The Protocol PI is the final arbiter of eligibility.
4. Subject has received a vaccination with a Live virus (e.g., Measles, Mumps, Rubella, Varicella).
5. Subject is pregnant or breastfeeding.
6. HIV seropositivity
7. Subjects who are unable to provide consent or who, in the opinion of the Investigator will be unlikely to fully comply with protocol requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-11 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Severe Infusion Toxicity as Assessed by CTCAE v4.0 | 24 hours post-intervention
  Number of Participants with Severe (Grade 3 or 4) Toxicity
Number of Participants with Regimen Related Death | 30 days post-intervention
  • severe (grade 3 or 4) cytokine release syndrome (CRS) within 30 days
Number of Participants with Severe Cytokine Release Syndrome (CRS) | 30 days post-intervention
  Number of Participants with Severe (Grade 3 or 4) CRS

CONTACTS AND LOCATIONS:
Overall Officials: Tara Sadeghi, Study Director — Sponsor GmbH

IPD SHARING:
Plan to Share IPD: No